CLINICAL TRIAL: NCT00806299
Title: An Open Label, Randomized, Single-dose, Fixed-Sequence Crossover Drug Interaction Study of Loperamide HCL With Grapefruit Juice
Brief Title: Loperamide Grapefruit Juice Interaction PK Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOPDIR1007
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Loperamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Drug (including placebo)
  Interventions: Drug: Loperamide / Red Grapefruit Juice
- 2 (Experimental): Drug (including placebo)
  Interventions: Drug: Loperamide/ White Grapefruit Juice
- 3 (Experimental): Drug (including placebo)
  Interventions: Drug: Loperamide / Pink Grapefruit Juice

INTERVENTIONS:
Drug: Loperamide / Red Grapefruit Juice — Fixed sequence of loperamide 4 mg with and without red grapefruit juice
  Other Names: Imodium
  Arms: 1
Drug: Loperamide/ White Grapefruit Juice — Fixed sequence of loperamide 4 mg with and without white grapefruit juice
  Other Names: Imodium
  Arms: 2
Drug: Loperamide / Pink Grapefruit Juice — Fixed sequence of loperamide 4 mg with and without pink grapefruit juice
  Other Names: Imodium
  Arms: 3

SUMMARY:
A 10-day study to determine if grapefruit juice has any effect on how loperamide (Imodium) affects the body and how the body affects loperamide.

DETAILED DESCRIPTION:
An open-label, randomized, single-dose, fixed-sequence crossover drug interaction study of loperamide HCl with grapefruit juice. About 33 healthy subjects, about equal numbers of men and women, 18 through 59 years of age, will be enrolled into this 10 day trial. Subjects will be divided into three cohorts of about 11 subjects each. Each cohort will receive red, white or pink grapefruit juice. Subjects will take 4 mg of loperamide on Day 1. They will ingest 8 ounces of grapefruit juice and then 4 mg of loperamide on Day 3. They will ingest 8 ounces of grapefruit juice in the morning and in the evening on Days 5, 6 and 7. On Day 8, subjects will ingest 8 ounces of juice and then 4 mg of loperamide. Blood samples will be collected at at predose (0) and 0.5, 1, 1.5, 32, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36 and 46 hours after dosing on Day 1, Day 3 and Day 8. Pupillometry assessments will be performed at pre-dose (0) and 2, 4, 6, 8, and 12 hours after dosing on Day 1, Day 3 and Day 8. Subjects will collect their urine from about 8 PM to about 6 AM prior to dosing on Day 1, Day 3 and Day 8.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 59 years, inclusive
* No clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, and clinical laboratory tests.
* Subjects will have a Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).
* Are normotensive with sitting blood pressure between the range of 90 - 140 mm Hg systolic and 50 - 90 mm Hg diastolic.
* Have a heart rate of 50-100 beats per minute (bpm).
* Have a negative urine drug screen at screening and at check-in to the research unit.
* If female of child-bearing potential, a negative pregnancy test at screening and at admission to the clinical research unit.
* Able to sign and date the informed consent document, indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Received a thorough explanation of the mandatory pharmacogenomic research component of the study and has signed the separate pharmacogenomic informed consent document.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Extensive restrictions on the type of food and drink allowed
* Medical history that precludes inclusion in the trial per protocol
* History of allergy and/or sensitivity to loperamide HCl
* History of alcohol consumption that precludes inclusion in the trial per protocol
* Positive screening test for HIV, Hepatitis B or Hepatitis C
* Treatment with an investigational drug within 30 days preceding the first dose of study medication
* Females who are pregnant, nursing, or unwilling or unable to use an acceptable method of nonhormonal contraception as outlined in the protocol
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives prior to first dose
* Donated or lost blood or blood products within 3 months of first dose or intention to donate blood or blood products within one month after the last dose
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Unwillingness or inability to comply with the Lifestyle Guidelines listed in the protocol
* Relationship to persons involved directly with the conduct of the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Blood samples will be collected before dosing (predose) and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 10, 14, 24, 30, 36, and 46 hours following each of the three doses

SECONDARY OUTCOMES:
Pharmacodynamic Parameter: Urine for Analysis of Cortisol and 6-beta Hydroxycortisol | 8 PM to about 6 AM prior to each dose administration, Day 1, Day 3 and Day 8
Pharmacodynamic Parameter: Pupillometry Assessments | predose (0) and at 2, 4, 6, 8, and 12 hours after dosing on Day 1, Day 3 and Day 8
Pharmacogenomic Evaluation - Genotype CYP3A4, CYP3A5, and ABCB1 | pre-dose or post-dose
Safety Assessments will consist of monitoring and recording all non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs), their frequency, severity, seriousness, and relationship to the investigational product | throughout duration of the study (+ 30 days for spontaneously reported SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Dolly Parasrampuria, PhD, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- Cetero Research, Fargo, North Dakota, United States